CLINICAL TRIAL: NCT06942403
Title: In-use Tolerance and Efficacy Study Under Dermatological Control of an Anti-aging Cream (Split Face) Post Facial Superficial Rejuvenation Procedures, After re Epidermization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RV4983A20230413
Record Dates: First submitted 2025-04-04; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: According to randomization, each subject will have a treated half face and a control half face.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treated group (hemiface) (Experimental)
  Interventions: Other: Associated product 1 : RV2666C; Other: Associated product 2 MORNING : RV5000A; Other: Test product : RV4983A
- Control group (hemiface) (Other)
  Interventions: Other: Associated product 1 : RV2666C; Other: Associated product 2 MORNING : RV5000A; Other: Associated product 2 EVENING: RV5000A

INTERVENTIONS:
Other: Associated product 1 : RV2666C — Applied twice a day minimum during 7 days (from Day 1 to Day 7)
Other: Associated product 2 MORNING : RV5000A — Applied in the mornings from Day 8 to Day 95 or Day 176*
  * for subjects post injections
Other: Test product : RV4983A — Applied once a day, at the evening. Avoid contact with eyes. If sensations of discomfort appear, allow more time between applications.
  * From Day 8 to Day 95 (87 days) for post LASER and post peeling subjects
  * From Day 8 to Day 176 (169 days) for post-injections subjects
  Arms: Treated group (hemiface)
Other: Associated product 2 EVENING: RV5000A — Applied in the evenings from Day 8 to Day 95 or Day 176*
  * for subjects post injections
  Arms: Control group (hemiface)

SUMMARY:
The aim of this study is to assess the dermatological tolerance of the investigational product "Crème visage Product code: RV4983A / Formula code: LA3365" after 95 days for subjects post peeling and LASER and 176 days for subjects post injections of once daily use at the evening on the half face, under normal conditions of use, on 66 subjects.

This study will be conducted as a national, monocentric, open trial.

Planning of the visits:

* Visit 1: Inclusion (Day 1) - The subjects undergo their procedure (peeling, LASER or injections).
* Home application of the associated product 1 period: Day 1 to Day 7
* Visit 2: intermediate visit (Day 8) subjects received investigational product and associated product 2;
* Visit 3, 4, and 5: Intermediate visit (Day 37, Day 66 and Day 95*),

  *the final visit for the subjects post peeling and LASER
* Visit 6**: End of study (Day 176), ** for subjects post injections

ELIGIBILITY:
Inclusion Criteria

Criteria related to the population:

* female and male
* aged between 35 and 70 years included
* phototype: I to IV
* all skin types
* subjects must be registered with health social security or health social insurance
* having signed their written Informed Consent form (ICF) for their participation in the study and a photograph authorization
* certifying the truth of the personal information declared to the Investigator able to understand the language used in the investigation centre and the information given
* able to comply with the protocol and follow protocol's constraints and specific requirements
* cooperative subject, aware of the necessity and duration of controls so that perfect adhesion to the protocol established by the clinical trial centre could be expected (able to comply with the protocol and follow protocol's constraints and specific requirements)
* a maximum of 20% of subjects being lens wearers will be included in the study

Criteria related to the skin condition:

- Subjects having performed superficial rejuvenation procedures on the face including the crow's foot area:

* 20 subjects after peeling (30 or 50% glycolic acid);
* 20 subjects after laser CO2
* 20 subjects after injections of hyaluronic acid or mix containing hyaluronic acid All procedures must remain superficial and aiming an anti-aging effect. Instrumental technics will be on the crow's foot so all procedures must be performed on the face including on this area.

Criteria related to subject's health:

* Considered "healthy subject" by the Investigator
* Women of childbearing potential committing themselves to use effective contraceptive method throughout the study and for at least 3 months before the inclusion visit (with no change during this period)

Non-Inclusion Criteria:

Criteria related to the population:

* having participated in another clinical trial within the week before the inclusion visit and for a longer period if required in the Investigator's opinion
* taking part or planning to participate in another clinical trial during the study in the same or another investigation centre
* breastfeeding, pregnant (for the women of childbearing potential)
* deprived of freedom by administrative or legal decision or under guardianship - not able to be contacted in case of emergency
* admitted in a sanitary or social facilities
* planning an hospitalization during the study
* belonging to the staff of the investigation centre

Criteria related to the skin condition

* having a dermatological condition liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
* having personal medical history liable to interfere with the study data for the subject or incompatible with the study requirements (except if this population is required by the Sponsor i.e atopic dermatitis)
* having history of abnormal reactions from exposure to sunlight
* having history of hypersensitivity or intolerance to any cosmetic product

Criteria related to treatments

* Topical or systemic treatment liable to interfere with the study data according to investigator's assessment
* having used a self-tanning product during the previous month
* having received, on the study areas, artificial UV exposure or excessive exposure to natural sunlight within the month before the inclusion visit (at Investigator's opinion)

Criteria related to investigational product application areas:

* having had any surgery, chemical or significant invasive dermo-treatment on the experimental area considered by the Investigator liable to interfere with the study data, before the inclusion visit or foreseeing it for the duration of the study (except if the treatment is required by the Sponsor)
* having applied a skincare or make up product on the study areas the day of the inclusion visit (except the usual cleanser)
* having received, on the study areas, artificial UV exposure or excessive exposure to natural sunlight within the 2 weeks before the inclusion visit

Criteria related to the COVID-19:

- subject who does not meet the Ministry of Health guidelines for Covid-19 at the time of the visit

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Assessment of dermatological physical signs by the investigator | At the Visit 2 (Day 8, before and immediately after investigational product application: 10 to 30 minutes) and at the Day 37, Day 66, Day 95 and Day 176 (for post-injections subjects) visit.
  The following signs are recorded by the investigator : erythema, oedema, desquamation, skin dry, vesicle, papule, any other sign observed.
  For each sign:
  * Intensity has to be reported by using the following scale: 0 none, 1 very mild, 2 mild, 3 moderate, 4 severe
  * For papules, vesicles, an estimation of the quantity is required instead of an intensity
  * Location, duration and frequency are also reported.
  Each time a sign occurs (either new sign or worsened compared to the baseline evaluation i.e evaluation at Day 8), a reaction is recorded in the CRF. Other signs present at the inclusion visit without any change in terms of severity are recorded as well in the CRF but not considered as reactions.
Assessment of dermatological functional signs by the subject | At the Visit 2 (Day 8, before and immediately after investigational product application: 10 to 30 minutes) and at the Day 37, Day 66, Day 95 and Day 176 (for post-injections subjects) visit
  The following signs are recorded by the subject : burning sensation, sensation of warmth, itching, skin tightness, stinging, any other sign observed.
  For each sign:
  * Intensity has to be reported by using the following scale: 0 none, 1 very mild, 2 mild, 3 moderate, 4 severe
  * Location, duration and frequency are also reported. Each time a sign occurs (either new sign or worsened compared to the baseline evaluation i.e evaluation at Day 8), a reaction is recorded in the CRF. Other signs present at the inclusion visit without any change in terms of severity are recorded as well in the CRF but not considered as reactions.
Recording of reactions | During the entire course of the study (from Day 1 to Day 95 or Day 176)
  All the reactions observed by the Investigator and reported by the subject are recorded.
  The following information are recorded:
  * Subject characteristics
  * Details about product
  * Description of the reaction
  * Significant medical history
  * Concomitant events
  * Outcome and actions taken
  * Relationship to the product (investigational product) : causality assessment The Investigator should assess the causality according to the three levels of causality : Very likely / Likely ; Not clearly attributable / Unlikely ; Excluded
Global tolerance assessment by the investigator | At the end of study (Day 176)
  Global tolerance will be assessed on the "tolerance population" which includes all the subjects who applied at least once investigational product.
  This assessment allows for attribution of one of the 5 levels below:
  * Excellent
  * Very good
  * Good
  * Moderate
  * Bad

SECONDARY OUTCOMES:
Smoothing/anti-wrinkle effect by instrumental measurements using 3D PRIMOS-LITE® | At the Visit 2 (Day 8, before investigational product application) and at the Day 37, Day 66, Day 95 and Day 176 (for post-injections subjects) visit.
Crow's feet wrinkles (according to Bazin scale) by the investigator | At the Visit 2 (Day 8, before and immediately after investigational product application: 10 to 30 minutes) and at the Day 37, Day 66, Day 95 and Day 176 (for post-injections subjects) visit.
Smoothness of the skin by the investigator | At the Visit 2 (Day 8, before and immediately after investigational product application: 10 to 30 minutes) and at the Day 37, Day 66, Day 95 and Day 176 (for post-injections subjects) visit.
  On a 11-points scale (0=wrinkled skin, 10=smooth skin)
Firmness of the skin by the investigator | At the Visit 2 (Day 8, before and immediately after investigational product application: 10 to 30 minutes) and at the Day 37, Day 66, Day 95 and Day 176 (for post-injections subjects) visit.
  On a 11-points scale (0=lack of firmness, 10=firm skin)
Skin plumpness by the investigator | At the Visit 2 (Day 8, before and immediately after investigational product application: 10 to 30 minutes) and at the Day 37, Day 66, Day 95 and Day 176 (for post-injections subjects) visit.
  On a 11-points scale (0=lack of plumpness, 10=plump skin)
Radiance of the complexion assessed by clinical scoring on pictures by technician | At the Visit 2 (Day 8, before investigational product application) and at the Day 37, Day 66, Day 95 and Day 176 (for post-injections subjects) visit.
  The complexion grading is performed on photographs (with Nikon®, in standard light) by a technician On a 11-points scale (0=Dull complexion, 10=radiant complexion)
Homogenity of skin tone assessed by clinical scoring on pictures by technician | At the Visit 2 (Day 8, before investigational product application) and at the Day 37, Day 66, Day 95 and Day 176 (for post-injections subjects) visit.
  The complexion grading is performed on photographs (with Nikon®, in standard light) by a technician On a 11-points scale (0=Not even at all, 10=very even skin texture)
Skin texture assessed by clinical scoring on pictures by technician | At the Visit 2 (Day 8, before investigational product application) and at the Day 37, Day 66, Day 95 and Day 176 (for post-injections subjects) visit.
  The complexion grading is performed on photographs (with Nikon®, in standard light) by a technician On a 11-points scale (0=Coarse, 10=Fine)
Visual expected effect | At the Visit 2 (Day 8, before investigational product application) and at the Day 37, Day 66, Day 95 and Day 176 (for post-injections subjects) visit.
  The device used is the VISIA® from CANFIELD® imaging systems. The VISIA allows taking pictures with multiple lighting modes and a very rapid capture of images. One photograph of the full face, each profile and crow feet is taken under multi-spectral imaging and analysis (normal light) allows capturing visual information
Cosmetic Acceptability evaluation by subjects | At the end of the study (Day 95 for post LASER and post peeling subjects, Day 176 for post injections subjects)
  A subjective evaluation questionnaire, prepared by the Sponsor, is filled in by the subjects at the end of the study to subjectively evaluate the properties, the efficacy, the tolerance and the future use of the studied product.
Subject's compliance regarding the test product recorded in their daily log checked by the investigator | During the entire course of the study (from Day 1 to Day 95 or Day 176)
  * Subjects are asked to keep a diary for recording of their daily applications details. This diary is returned by the subject at each visit to be checked by the investigator
  * A compliant subject will be defined as a subject who did apply the investigational product sufficiently to not interfere with the study data according to the Investigator's opinion and the modalities of use of the product.
  * List of non-compliant subjects will be displayed in the study report.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermscan Poland, Gdansk, Poland, Poland

REFERENCES:
- [Derived] Monteil C, Barreto-Campos V, Lain E, Guillou E, Doat G, Nocera T. Enhancing Facial Rejuvenation Outcomes With a Novel Retinaldehyde-Based Cream: A Comparative Randomized Intra-Individual Study. J Cosmet Dermatol. 2025 Dec;24(12):e70555. doi: 10.1111/jocd.70555. PMID 41312593